CLINICAL TRIAL: NCT05801224
Title: Regional Vascular Recruitment With Inhaled Nitric Oxide in Patients With ARDS
Brief Title: Vascular ARDS Recruitment After Inhaled Nitric Oxide
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is now funded by NIH grant R01HL171199, and recruitment is planned to start in July 2026 per the grant timeline.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Maurizio F. Cereda, MD, MD, Member of the Faculty of Anaesthesia, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023p000138
Record Dates: First submitted 2023-03-11; First posted 2023-04-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Distress Syndrome; Ventilation Perfusion Mismatch
Keywords: Acute respiratory distress syndrome; Ventilation/perfusion mismatch; Electrical impedance tomography; Inhaled nitric oxide; Dual-energy computed tomography
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Intervention Model Description: In a prospective, single-center, physiological, crossover study, the investigators will recruit 70 adults meeting the ARDS criteria based on the Berlin definition who have not previously received inhaled vasodilators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Electrical Impedance Tomography (Experimental): A total of 60 subjects (cohort 1) will receive an inhaled nitric oxide (iNO) challenge (20 ppm) for 15 min. The investigators will measure ventilation and perfusion distributions using EIT before iNO ("OFF1"), after 15 min on iNO ("ON"), and after 15 min washout ("OFF2") to confirm baseline stability.
  Interventions: Device: Nitric Oxide
- Electrical Impedance Tomography and Dual-Energy Computed Tomography (Experimental): In a subset of 10 subjects (cohort 2), EIT and DECT will be performed in a row at the same type of bed and body position. In cohort 2, the measurements will be before nitric oxide (iNO) and during iNO. The OFF-ON fashion for DECT imaging is to minimize the subject's exposure to radiation and reduce the time spent in the CT room.
  Interventions: Device: Nitric Oxide

INTERVENTIONS:
Device: Nitric Oxide — 20ppm for 15 minutes delivered by INO max(Nitric Oxide) Company : INO therapeutics, Inc.
  Other Names: inhaled nitric oxide (iNO)

SUMMARY:
Acute respiratory distress syndrome (ARDS) is when a person's lungs become inflamed, which can be caused by infection, trauma, surgery, blood transfusion, or burn. ARDS often leads to a situation where the person cannot breathe independently and needs machines' help. Once the lungs are inflamed, the small air sacs responsible for exchanging gases (i.e., ventilation) and the blood flow in the lungs (i.e., perfusion) can be affected. In the past, most research focused on studying ventilation physiology and how to help people breathe with machines. Less was done on perfusion because it requires imaging techniques such as computed tomography with intravenous contrast and radiation. One treatment option for low oxygen levels is inhaled nitric oxide (iNO), a gas that can dilate the lung blood vessels and improve oxygenation; however, it is not always clear whether this treatment will work. Electrical Impedance Tomography (EIT) is a bedside and accessible imaging technique that is radiation-free and non-invasive and can potentially detect changes in lung perfusion. EIT can perform multiple measurements; it is portable and accessible. This prospective interventional study aims to assess changes in regional blood perfusion in the lungs of patients with ARDS in response to iNO utilizing EIT. The main questions it aims to answer are:

1. If EIT can measure lung regional perfusion response to an iNO challenge of 20ppm for 15 minutes.
2. If EIT is comparable to dual-energy computed tomography (DECT), the gold-standard method to detect changes in regional lung perfusion.
3. If EIT can be an imaging marker to identify ARDS severity

Participants will be divided into two cohorts:

1. Cohort 1 (n=60): Participants will be asked to be monitored by EIT before, during, and after the administration of iNO (20 ppm) for 15 minutes (OFF-ON-OFF)
2. Cohort 2 (N=10): Participants will be asked to be monitored by EIT and DECT before and during the administration of iNO (20 ppm) for 15 minutes (OFF-ON).

DETAILED DESCRIPTION:
The investigators will screen patients with ARDS diagnosis daily at MGH intensive care units and work in the consenting process with the ICU team and surrogates. The enrollment period will be limited to the time subjects will undergo the study procedures. Subjects will exit the study as soon as the study procedures are completed. No further procedures are planned; therefore, subjects will not be asked to return to the hospital exclusively for research-related purposes.

The enrolled subjects will be divided into two cohorts. Cohort 1 (n=60) will be monitored with EIT before, during, and after the administration of iNO. Cohort 2 (n=10) will be monitored with EIT and DECT before and during the administration of iNO.

Methods to answer question 1 (To measure the topographic perfusion response to an iNO challenge with EIT):

- The EIT monitoring will be composed of ventilation and perfusion distributions. First, the ventilation is recorded; at this point, no additional maneuver is needed; the subjects need to wear the electrode belt connected to the device, and their ventilation will be recorded. Secondly, for the perfusion distribution, after a pause in the ventilation, EIT measures the distribution of blood perfusion in the lungs during the injection of a 10 mL bolus of 11.7% hypertonic saline solution through a central venous catheter. Cohort 1 (n=60) will receive 20ppm of iNO for 15 minutes. Cohort 1 will be monitored with EIT before, during, and after the iNO delivery in an OFF-ON-OFF fashion.

Methods to answer question 2 (To compare EIT measurements against the gold standard DECT):

- Cohort 2 (n=10) will be monitored with EIT and DECT. They will receive 20ppm of iNO for 15 minutes. The subjects will be transported to the computed tomography (CT) room, and the first DECT (DECT OFF) will be performed before the iNO delivery. After the DECT OFF, the EIT belt will be placed, and ventilation/perfusion will be measured before the iNO delivery (EIT OFF). Then, the iNO delivery will start, and after 15 minutes, the EIT ON will be recorded. The EIT belts will be removed, and the second DECT (DECT ON) will be performed. Of note, the EIT belt needs to be removed before the DECT acquisitions because the electrodes generate artifacts that would compromise the image quality.

Methods to answer question 3 (To determine ARDS phenotypes based on regional perfusion imaging):

- The investigators will explore the vascular response measured by EIT and categorize subjects accordingly. The investigators plan to apply EIT patterns as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.

Finally,

* Blood MetHb levels will be continuously monitored before, during, and after each iNO administration of the day. At the end of each iNO administration, MetHb will continue to be monitored until values return to the level recorded before the current treatment and
* The NO, nitrogen dioxide (NO2) will be continuously monitored by INOmax DSIR (Mallinckrodt) deliver system.

ELIGIBILITY:
Inclusion Criteria:

* Adult intubated and mechanically ventilated patients (≥ 18 years old) admitted to the intensive care unit (ICU)
* ARDS diagnosis with mild to moderate severity by Berlin criteria1 (100 mmHg < PaO2/FiO2 <= 300 mmHg)
* Presence of an arterial line for blood gas measurement and blood pressure monitoring and of a central line for hypertonic saline injection

Exclusion Criteria:

* Suspected pregnancy, pregnancy or less than six weeks postpartum
* Younger than 18 years or older than 80 years
* Baseline methemoglobin ≥ 5%
* Subjects enrolled in another interventional research study
* Presence of pneumothorax
* Usage of any devices with electric current generation, such as a pacemaker or internal cardiac defibrillator
* Preexisting chronic lung disease or pulmonary hypertension
* Past medical history of lung malignancy or pneumonectomy, or lung transplant
* Left ventricle ejection fraction <20%
* Hemodynamic instability is defined as:

  * Persistent systolic blood pressure <90 mmHg and/or >180 mmHg despite the use of vasopressor or vasodilators, or
  * Requiring an increment in inotropic vasopressors over the past two hours just before enrollment: more than 15 mcg/min for norepinephrine and dopamine, more than 10 mcg/min in epinephrine, and more than 50 mcg/ min for phenylephrine.
* Hypernatremia (serum sodium > 150 mEq/L)
* Patients cannot be enrolled for DECT if they have:

  * History of allergic reaction to intravenous contrast
  * Renal dysfunction on the day of the study (serum creatinine > 1.5 mg/dL)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in regional lung perfusion after the delivery of inhaled nitric oxide | Day 1
  The primary outcome is to detect changes in regional perfusion distribution with the administration of inhaled nitric oxide with electrical impedance tomography by measuring changes in impedance.

SECONDARY OUTCOMES:
Compare methods to detect change in regional lung perfusion after the delivery of inhaled nitric oxide | Day 1
  The secondary outcome is to To compare electrical impedance tomography measurements against the gold standard dual-energy computed tomography (DECT)

OTHER OUTCOMES:
Age | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
  Age (years)
Gender | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Height | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Weight | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Race | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Ethnicity | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Comorbidities | Day 1
  Presence in the past medical history of conditions such as hypertension, diabetes,obesity, COPD, liver disease, and heart failure, among others.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Hours Elapsed since intubation | Day 1
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Apache II score | Within 24 hours of intensive care admission
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Intensive care unit survival at 28 days | Day 28
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Hospital survival at 28 days | Day 28
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Ventilation-free days | From day 1 to day 28
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
PaO2 | Day 1, arterial blood gas samples will be taken at two time points: before and 1 hour after iNO. Subsequent days up to 28 days will be determined by the critical care staff
  The PaO2 will be measured with an arterial blood sample. This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
PaCO2 | Day 1, arterial blood gas samples will be taken at two time points: before and 1 hour after iNO. Subsequent days up to 28 days will be determined by the critical care staff
  The PaCO2 will be measured with an arterial blood sample. This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Ph | Day 1, arterial blood gas samples will be taken at two time points: before and 1 hour after iNO. Subsequent days up to 28 days will be determined by the critical care staff
  The Ph will be measured with an arterial blood sample. This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Methemoglobin (MetHb) | Day 1, arterial blood gas samples will be taken at two time points: before and 1 hour after iNO. Subsequent days up to 28 days will be determined by the critical care staff
  The MetHb will be measured with an arterial blood sample. This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
HCO3 (bicarbonate) | Day 1, arterial blood gas samples will be taken at two time points: before and 1 hour after iNO. Subsequent days up to 28 days will be determined by the critical care staff
  The HCO3 will be measured with an arterial blood sample. This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Tidal Volume | From day 1 to day 28
  Ventilator Parameter. This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Plateau, peak and positive end-expiratory pressures | From day 1 to day 28
  Ventilator Parameters are measured during tidal ventilation, inspiratory and expiratory holds.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Respiratory rate | From day 1 to day 28
  Ventilator Parameters are measured during tidal ventilation, inspiratory and expiratory holds.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Flow | From day 1 to day 28
  Ventilator Parameters are measured during tidal ventilation, inspiratory and expiratory holds.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Vasopressors requirements (dopamine, dobutamine, epinephrine, levosimendan, milrinone, vasopressin, norepinephrine) | From day 1 to day 28
  We will calculate the Vasoactive-inotropic score (VIS). The VIS compares different vasoactive-inotropic drugs and doses among the patients.
  VIS = dopamine dose (mg/kg/min)+ dobutamine [mg/kg/min) +100 x epinephrine dose (mg/ kg/min) +50 x levosimendan dose [mg/kg/min) + 10 x milrinone dose [mg/kg/min)+ 10,000 x vasopressin [units/kg/min) + 100x norepinephrine dose [mg/kg/min) using the maximum dosing rates of vasoactive and inotropic medications.
  Ref: Koponen et al. British Journal of Anaesthesia, 122 (4): 428e436 (2019).
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Arterial blood pressure, central venous pressure, pulmonary artery pressure | From day 1 to day 28
  Hemodynamic parameters. The pulmonary artery pressure will be measured if the subject have a pulmonary artery pressure placed by the ICU staff with clinical purposes.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
Life sustaining therapies | From day 1 to day 28
  Other life-sustaining therapies than mechanical ventilation and vasopressors administration: Antibiotics, Renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO), chemotherapy, and artificial nutrition.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.
CRP, MCP-1, TNF-alpha, IL-6, IL-8, IL-10, Ang-2, VEGF | From day 1 to day 28
  Blood samples will be collected and Systemic markers of inflammation and plasma cytokines: CRP, MCP-1, TNF-alpha, IL-6, IL-8, IL-10, Ang-2, VEGF will be measured.
  This exploratory outcome plans to utilize electrical impedance tomography as an image marker and combine them with other markers (demographical, radiological, clinical, biochemical, and inflammatory) to identify ARDS sub-phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Cereda, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Matthay MA, Zemans RL, Zimmerman GA, Arabi YM, Beitler JR, Mercat A, Herridge M, Randolph AG, Calfee CS. Acute respiratory distress syndrome. Nat Rev Dis Primers. 2019 Mar 14;5(1):18. doi: 10.1038/s41572-019-0069-0. PMID 30872586
- [Background] Cressoni M, Caironi P, Polli F, Carlesso E, Chiumello D, Cadringher P, Quintel M, Ranieri VM, Bugedo G, Gattinoni L. Anatomical and functional intrapulmonary shunt in acute respiratory distress syndrome. Crit Care Med. 2008 Mar;36(3):669-75. doi: 10.1097/01.CCM.0000300276.12074.E1. PMID 18091555
- [Background] Zapol WM, Kobayashi K, Snider MT, Greene R, Laver MB. Vascular obstruction causes pulmonary hypertension in severe acute respiratory failure. Chest. 1977 Feb;71(2 suppl):306-7. doi: 10.1378/chest.71.2_supplement.306. No abstract available. PMID 836381
- [Background] Greene R, Zapol WM, Snider MT, Reid L, Snow R, O'Connell RS, Novelline RA. Early bedside detection of pulmonary vascular occlusion during acute respiratory failure. Am Rev Respir Dis. 1981 Nov;124(5):593-601. doi: 10.1164/arrd.1981.124.5.593. No abstract available. PMID 7305115
- [Background] Tomashefski JF Jr, Davies P, Boggis C, Greene R, Zapol WM, Reid LM. The pulmonary vascular lesions of the adult respiratory distress syndrome. Am J Pathol. 1983 Jul;112(1):112-26. PMID 6859225
- [Background] Rossaint R, Falke KJ, Lopez F, Slama K, Pison U, Zapol WM. Inhaled nitric oxide for the adult respiratory distress syndrome. N Engl J Med. 1993 Feb 11;328(6):399-405. doi: 10.1056/NEJM199302113280605. PMID 8357359
- [Background] Johnson TR. Dual-energy CT: general principles. AJR Am J Roentgenol. 2012 Nov;199(5 Suppl):S3-8. doi: 10.2214/AJR.12.9116. PMID 23097165
- [Background] Borges JB, Suarez-Sipmann F, Bohm SH, Tusman G, Melo A, Maripuu E, Sandstrom M, Park M, Costa EL, Hedenstierna G, Amato M. Regional lung perfusion estimated by electrical impedance tomography in a piglet model of lung collapse. J Appl Physiol (1985). 2012 Jan;112(1):225-36. doi: 10.1152/japplphysiol.01090.2010. Epub 2011 Sep 29. PMID 21960654
- [Result] Safaee Fakhr B, Araujo Morais CC, De Santis Santiago RR, Di Fenza R, Gibson LE, Restrepo PA, Chang MG, Bittner EA, Pinciroli R, Fintelmann FJ, Kacmarek RM, Berra L. Bedside monitoring of lung perfusion by electrical impedance tomography in the time of COVID-19. Br J Anaesth. 2020 Nov;125(5):e434-e436. doi: 10.1016/j.bja.2020.08.001. Epub 2020 Aug 7. No abstract available. PMID 32859359
- [Result] Morais CCA, Safaee Fakhr B, De Santis Santiago RR, Di Fenza R, Marutani E, Gianni S, Pinciroli R, Kacmarek RM, Berra L. Bedside Electrical Impedance Tomography Unveils Respiratory "Chimera" in COVID-19. Am J Respir Crit Care Med. 2021 Jan 1;203(1):120-121. doi: 10.1164/rccm.202005-1801IM. No abstract available. PMID 33196303
- [Result] De Santis Santiago R, Teggia Droghi M, Fumagalli J, Marrazzo F, Florio G, Grassi LG, Gomes S, Morais CCA, Ramos OPS, Bottiroli M, Pinciroli R, Imber DA, Bagchi A, Shelton K, Sonny A, Bittner EA, Amato MBP, Kacmarek RM, Berra L; Lung Rescue Team Investigators. High Pleural Pressure Prevents Alveolar Overdistension and Hemodynamic Collapse in Acute Respiratory Distress Syndrome with Class III Obesity. A Clinical Trial. Am J Respir Crit Care Med. 2021 Mar 1;203(5):575-584. doi: 10.1164/rccm.201909-1687OC. PMID 32876469